CLINICAL TRIAL: NCT05437549
Title: CMR Characterization of Ablation Lesions Following Pulmonary Vein Isolation
Brief Title: Evaluating PVI Using CMR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, Luuk Hopman, PhD student, Amsterdam UMC, location VUmc
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NL75456.029.20
Record Dates: First submitted 2022-06-17; First posted 2022-06-29 (Actual); Last update posted 2022-06-29 (Actual); Status verified 2022-06

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PVI (Other)
  Interventions: Procedure: MRI

INTERVENTIONS:
Procedure: MRI — MRI prior to PVI, acutely after PVI, and 3 months after PVI

SUMMARY:
Using state of the art cardiac magnetic resonance imaging techniques, characterization of ablation lesions in the early phase after pulmonary vein isolation ablation in atrial fibrillation patients, and relate findings to the ablation scar at 3 months follow up and atrial fibrillation-free survival at 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age ≥18 years old)
* Paroxysmal or persistent AF meeting guideline criteria.
* Anticipated PVI using index-guided radiofrequency ablation techniques.
* Availability of LGE-CMR images within 3 months before anticipated PVI.

Exclusion Criteria:

* History of catheter ablation
* History of cardiac surgery.
* History of chest radiation therapy
* Estimated glomerular filtration rate (eGFR) <45 ml/min/kg
* Known (or suspected) allergic reaction to gadolinium
* Contraindications for CMR (such as claustrophobia, certain implants, devices, high body mass index).
* Inability to schedule CMR <48h after PVI
* Long-term use of anti-inflammatory medication, except for the use of nonsteroidal anti-inflammatory drugs
* Autoimmune disease or chronic inflammatory illness.
* Pregnancy of breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Ablaton scar | 3 months
  The correlation between ablation lesion characteristics in the early phase after PVI and ablation scar at 3 months follow up.

SECONDARY OUTCOMES:
AF recurrence | 1 year
  The relation between ablation lesion characteristics and AF recurrence at 1 year after the ablation procedure